CLINICAL TRIAL: NCT03935698
Title: Physiotherapy Treatment in Gynecological Cancer Survivors Suffering From Dyspareunia: a Mixed-Method Pilot Study
Brief Title: Physiotherapy Treatment in Women With Dyspareunia Following Gynecological Cancer: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Institut Universitaire de Gériatrie de Montréal (Other); Jewish General Hospital (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Mélanie Morin, Researcher and Associate Professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-31-2016-1322
Record Dates: First submitted 2019-04-10; First posted 2019-05-02 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Gynecological Cancer; Dyspareunia
Keywords: Pilot study; Feasibility study; Dyspareunia; Gynecological cancer survivors; Physiotherapy
MeSH Terms: conditions — Dyspareunia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Pre-treatment assessment - Intervention (12 weeks) - Post-treatment assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy (Experimental): 12 weekly 60-minute individual sessions of multimodal physiotherapy including education, stretching techniques, pelvic floor muscle biofeedback as well as home exercises.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy
  Other Names: Pelvic floor rehabilitation

SUMMARY:
Gynecological cancers represent more than half of female cancers. It has been clearly established that cancer survivors suffer from important health issues such as pain during sexual intercourse (dyspareunia) and sexual dysfunctions which sorely impact their quality of life. Although it affects more than 63% of cancer survivors, the available treatments remain limited and poorly studied. Cancer survivors are thus confronted with these health issues as well as relationship difficulties and psychological consequences, with limited treatment avenues. Addressing pelvic floor muscle dysfunctions and loss of vaginal elasticity, pelvic floor physiotherapy was shown to be effective in reducing or even alleviating dyspareunia and improving sexual function. Until now, no study investigated this treatment in gynecological cancer survivors with dyspareunia. Therefore, there is a need to examine pelvic floor physiotherapy to determine whether or not gynecological cancer survivors with dyspareunia could benefit from this treatment. The objectives of this single-arm mixed-method study are to evaluate the acceptability and feasibility of a physiotherapy treatment in gynecological cancer survivors suffering from dyspareunia and to explore treatment effects. This single-arm study using mixed methods will involve three data collections (pre- and post-treatment assessments). These assessments will be carried out by physiotherapists. Participants will receive physiotherapy treatment weekly in individual 60-minute sessions for 12 weeks. Thirty-one gynecological cancer survivors with vulvovaginal pain during sexual intercourse for at least 3 months will be recruited. The results of this study will bring new information regarding physiotherapy treatment for this population in preparation for a definitive randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* History of gynecological cancer (endometrial, cervical, vaginal or other parts of the uterus)
* Scheduled oncological treatments completed with no signs of cancer for at least 3 months
* Vulvovaginal pain during sexual intercourse for at least 3 months

Exclusion Criteria:

* Vulvovaginal pain before cancer and not related to sexual intercourse
* Medication recognized to affect pain
* Refuse to stop other treatments until post-treatment assessment
* Other conditions interfering with assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Adherence rates | Pre- to 2-week post-treatment assessment
  To determine acceptability.
Retention rate | Pre- to 2-week post-treatment assessment
  To determine feasibility.

SECONDARY OUTCOMES:
Change from baseline in pain | Pre- to 2-week post-treatment assessment
  To explore changes in pain during sexual intercourse (Numerical Rating Scale, ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever).
Change from baseline in sexual function | Pre- to 2-week post-treatment assessment
  To explore changes in sexual function (Female Sexual Function Index).
Change from baseline in pelvic floor muscle function | Pre- to 2-week post-treatment assessment
  To explore changes in pelvic floor muscle function at rest and during contraction (dynamometry and ultrasound).
Change from baseline in quality of life | Pre- to 2-week post-treatment assessment
  To explore changes in quality of life (questionnaire).
Patient's global impression of change | 2-week post-treatment assessment
  To determine patient self-reported improvement (Patient's Global Impression of Change).
Adverse events | Pre- to 2-week post-treatment assessment
  To document any adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche du Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cyr MP, Dumoulin C, Bessette P, Pina A, Gotlieb WH, Lapointe-Milot K, Mayrand MH, Morin M. Changes in pelvic floor morphometry and muscle function after multimodal physiotherapy for gynaecological cancer survivors suffering from dyspareunia: a prospective interventional study. Physiotherapy. 2022 Mar;114:54-62. doi: 10.1016/j.physio.2021.09.003. Epub 2021 Sep 30. PMID 35093737